CLINICAL TRIAL: NCT03300973
Title: Role of Urodynamic Study Before Surgery for Stress Urinary Incontinence.
Brief Title: Urodynamic Study and Stress Incontinence
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Kasr El Aini Hospital (Other)
Responsible Party: Principal Investigator, sarah mohamed hassan, lecturer of obstetrics and gynecology Cairo university, Kasr El Aini Hospital
Allocation: Randomized | Model: Parallel | Purpose: Treatment
Other Study IDs: 11279
Record Dates: First submitted 2017-09-21; First posted 2017-10-04 (Actual); Last update posted 2017-10-04 (Actual); Status verified 2017-09

CONDITIONS: Stress Urinary Incontinence
Keywords: urodynamic study; stress urinary incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- urodynamics study group (Active Comparator): 65 patients with stress urinary incontinence were randomly chosen to have urodynamic study before surgery
  Interventions: Procedure: sling surgery
- surgery only group (Active Comparator): 60 patients with stress urinary incontinence were randomly chosen to have surgery without urodynamics study
  Interventions: Procedure: sling surgery

INTERVENTIONS:
Procedure: sling surgery — transoburator vaginal tape ,inside out procedure under spinal anathesia

SUMMARY:
A trial to answer the debatabal question about the role of urodynamic study in surgical treatment for stress urinary incontinence.

DETAILED DESCRIPTION:
group of patients complaining of stress urinary incontinence and candidate for sling surgery were randomaly divided into 2 groups either to have urodynamic study before surgery or not.

ELIGIBILITY:
Inclusion Criteria:

* stress urinary incontinence

Exclusion Criteria:

* mixed incontinence
* recurrent cases

Ages: 20 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 125 (Estimated)
Dates: Start 2016-01-15 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
cure of stress incontinence | 1 week after surgery
  by clinical assessment

SECONDARY OUTCOMES:
cure of stress incontinence | one month after surgery
  by clinical assessment
cure of stress incontinence | 3 months after surgery
  by clinical assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr El Ainiy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No